CLINICAL TRIAL: NCT00995137
Title: Pilot Study of Genetically Modified Haploidentical Natural Killer Cell Infusions for B-Lineage Acute Lymphoblastic Leukemia
Brief Title: Genetically Modified Haploidentical Natural Killer Cell Infusions for B-Lineage Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Assisi Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKCD19; R01CA113482 (NIH); NCI-2011-01226 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2015-02

CONDITIONS: Lymphoblastic Leukemia, Acute
Keywords: Relapsed or refractory B-Lineage ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- relapse B-Lineage ALL (Experimental): All patients meeting the eligibility criteria.
  Intervention: NK Cell Infusion
  Interventions: Biological: NK Cell Infusion

INTERVENTIONS:
Biological: NK Cell Infusion — Infusing genetically modified NK cells into research participants who have chemotherapy refractory or relapse B-lineage ALL.

SUMMARY:
This study will determine the maximum tolerated dose of genetically modified natural killer (NK) cells in research participants with relapsed or refractory B-lineage acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
NK cell cytotoxicity is most powerful against acute myeloid leukemia (AML) cells, whereas their capacity to lyse ALL cells is generally low and difficult to predict. A novel method has been developed to redirect NK cells towards CD19, a molecule highly expressed on the surface of B-lineage ALL cells, but not expressed on normal cells other than B-lymphocytes. In this method, donor NK cells are first expanded by co-culture with irradiated K562 cell line modified to express membrane bound IL-15 and 41BB ligand (K562-mb15-41BBL). Overexpansion of these proteins promotes selective growth of NK cells. Then, the expanded NK cells are transduced with a signaling receptor that binds to CD19 (anti-CD19-BB-zeta). NK cells expressing these receptors showed powerful anti-leukemic activity against CD19+ ALL cells in vitro and in an animal model of leukemia.

This study represents the translation of laboratory findings into clinical application. It will allow us to assess the safety of infusing genetically modified NK cells into research participants who have chemotherapy refractory or relapse B-lineage ALL. In this same cohort, we also intend to study the in vivo lifespan and phenotype of genetically modified NK cells and explore the efficacy of NK cells in patients with B-lineage ALL.

ELIGIBILITY:
Inclusion Criteria:

* Age: less than or equal to 18 years of age. May be greater than 18 years of age if currently a St. Jude patient.
* Patients with relapsed or refractory B-lineage ALL who are not eligible for hematopoietic stem cell transplantation (HSCT) because their leukemia is not in remission (>5% blasts in bone marrow as evidenced either by morphology or by flow cytometry).
* Shortening fraction greater than or equal to 25%.
* Glomerular filtration rate greater than or equal to 50 cc/min/1.73 m2.
* Pulse oximetry greater than or equal to 92% on room air.
* Direct bilirubin less than or equal to 3.0 mg/dL.
* Alanine aminotransferase (ALT) is no more than 2 times the upper limit of normal.
* Aspartate transaminases (AST) is no more than 2 times the upper limit of normal.
* Karnofsky or Lansky performance score of greater than or equal to 50.
* No known allergy to murine products or HAMA testing results within normal limits.
* No prior receipt of a gene-transfer agent (e.g. retroviral, adenoviral, lentiviral vector).
* Does not have a current pleural or pericardial effusion.
* Has a suitable adult family member donor available for NK cell donation.
* Has recovered from all acute NCI Common Toxicity Criteria grade II-IV non-hematologic acute toxicities resulting from previous therapy as per the judgment of the principal investigator.
* At least two weeks since receipt of any biological therapy, systemic chemotherapy, and/or radiation therapy.
* Is not receiving more than the equivalent of prednisone 10 mg daily.

Exclusion Criteria:

* Pregnant (negative serum or urine pregnancy test to be conducted within 7 days prior to enrollment)
* Breastfeeding

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2009-10; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
This study will determine the maximum tolerated dose of genetically modified NK cells in research participants with relapsed or refractory B-lineage ALL | 30 days after the enrollment of the last patient

SECONDARY OUTCOMES:
This study will determine the persistence and phenotype of genetically modified NK cells in research participants with relapsed or refractory B-lineage ALL. | 30 days after the enrollment of the last patient
This study will explore the efficacy of genetically modified NK cells in research participants with relapsed or refractory B-lineage ALL. | 30 days after the enrollment of the last patient

CONTACTS AND LOCATIONS:
Overall Officials: David Shook, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Del Zotto G, Marcenaro E, Vacca P, Sivori S, Pende D, Della Chiesa M, Moretta F, Ingegnere T, Mingari MC, Moretta A, Moretta L. Markers and function of human NK cells in normal and pathological conditions. Cytometry B Clin Cytom. 2017 Mar;92(2):100-114. doi: 10.1002/cyto.b.21508. Epub 2017 Feb 12. PMID 28054442
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols